CLINICAL TRIAL: NCT01848028
Title: Long-Term Benefits and Safety of Systemic Psoriasis Therapy: German Registry on the Treatment of Psoriasis With Biologics and Systemic Therapeutics
Brief Title: PsoBest - The German Psoriasis Registry
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Berufsverband der Deutschen Dermatologen e.V. (www.bvdd.de) (Unknown); Deutsche Dermatologische Gesellschaft e.V. (https://derma.de) (Unknown); AbbVie (Industry); Biogen (Industry); Janssen-Cilag G.m.b.H (Industry); medac GmbH (Industry); Merck Sharp & Dohme LLC (Industry); Novartis Pharmaceuticals (Industry); Pfizer Pharmaceuticals Ltd. (Industry); Merck Serono GmbH, Germany (Industry); PsoNet.eu (http://www.psonet.eu/) (Unknown); Celgene (Industry); Eli Lilly and Company (Industry); Amgen (Industry); Almirall Hermal GmbH (Industry); UCB Pharma (Industry); Bristol-Myers Squibb (Industry); Viatris Inc. (Industry); LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: IVDP-085-07
Record Dates: First submitted 2013-04-07; First posted 2013-05-07 (Estimated); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Psoriasis; Psoriatic-arthritis
Keywords: patient registry; Germany; psoriasis; psoriatic-arthritis; biologics; Psonet; effectiveness; safety; biosimilars
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (25):
- Fumaric acid esters: Intervention: Drug: conventional systemic: Fumaric acid esters, including Dimethylfumarate, all dosages, frequencies and durations prescribed
- Methotrexate: Intervention: Drug: conventional systemic: Methotrexate, all dosages, frequencies and durations prescribed
- Cyclosporine A: Intervention: Drug: conventional systemic: Cyclosporine A, all dosages, frequencies and durations prescribed
- Efalizumab (withdrawn): Intervention: Biological: Efalizumab, all dosages, frequencies and durations prescribed
- Etanercept: Intervention: Biological and biosimilars: Etanercept, all dosages, frequencies and durations prescribed
- Infliximab: Intervention: Biological and Biosimilars/-identicals: Infliximab, all dosages, frequencies and durations prescribed
- Adalimumab: Intervention: Biological and Biosimilars: Adalimumab, all dosages, frequencies and durations prescribed
- Ustekinumab: Intervention: Biological and Biosimilars: Ustekinumab, all dosages, frequencies and durations prescribed
- Golimumab: Intervention: Biological: Golimumab, all dosages, frequencies and durations prescribed
- Secukinumab: Intervention: Biological: Secukinumab, all dosages, frequencies and durations prescribed
- Apremilast: Intervention: Small molecule: Apremilast, all dosages, frequencies and durations prescribed
- Certolizumab: Intervention: Biological: Certolizumab, all dosages, frequencies and durations prescribed
- Retinoids: Intervention: Drug: conventional systemic: Retinoids, all dosages, frequencies and durations prescribed
- Leflunomids: Intervention: Drug: conventional systemic: Leflunomids, all dosages, frequencies and durations prescribed
- systemic PUVA: Intervention: Drug: conventional systemic: systemic PUVA, all dosages, frequencies and durations prescribed
- Guselkumab: Intervention: Biological: Guselkumab all dosages, frequencies and durations prescribed
- Brodalumab: Intervention: Biological: Brodalumab, all dosages, frequencies and durations prescribed
- Tildrakizumab: Intervention: Biological: Tildrakizumab, all dosages, frequencies and durations prescribed
- Risankizumab: Intervention: Biological: systemic Risankizumab, all dosages, frequencies and durations prescribed
- Bimekizumab: Intervention: Biological: Bimekizumab, all dosages, frequencies and durations prescribed
- Tofacitinib: Intervention: JAK-Inhibitor: Tofacitinib, all dosages, frequencies and durations prescribed
- Upadacitinib: Intervention: JAK-Inhibitor: Upadacitinib, all dosages, frequencies and durations prescribed
- Deucravacitinib: Intervention: JAK-Inhibitor: Deucravacitinib, all dosages, frequencies and durations prescribed
- Ixekizumab: Intervention: Biological: Ixekizumab, all dosages, frequencies and durations prescribed
- No treatment: Intervention: no systemic treatment in observation episodes

SUMMARY:
Treatment of moderate to severe Psoriasis (Pso) and Psoriasis-Arthritis (PsA) is largely confined to systemic therapy in Germany. Systemic therapy includes conventional systemic therapy (e.g. fumaric acids, methotrexate, ciclosporin A) and biological treatment (e.g. adalimumab, etanercept). While short- and middle-term efficacy of most systemic treatments has been shown in clinical studies (and is incorporated in international guidelines), knowledge about long-term outcomes, optimal treatment and effectiveness under real-world conditions is still missing. PsoBest, the German registry on the treatment of moderate to severe Pso and PsA started in 2008 and documents the long-term course of patients being administered any biologic or conventional systemic antipsoriatic drug authorized in Germany for the first time. The registry evaluates the long-term course of 3,500 patients with Pso and PsA treated with systemic antipsoriatics.

DETAILED DESCRIPTION:
Background: Treatment of moderate to severe Psoriasis (Pso) and Psoriasis-Arthritis (PsA) is largely confined to systemic therapy in Germany. Systemic therapy includes conventional systemic therapy (e.g. fumaric acids, methotrexate, ciclosporin A) and biological treatment (e.g. adalimumab, etanercept). While short- and middle-term efficacy of most systemic treatments has been shown in clinical studies (and is incorporated in international guidelines), knowledge about long-term outcomes, optimal treatment and effectiveness under real-world conditions is still missing. PsoBest, the German registry on the treatment of moderate to severe Pso and PsA started in 2008 and documents the long-term course of patients being administered any biologic or conventional systemic antipsoriatic drug authorized in Germany for the first time.

Objectives: Observation and analysis of the following outcomes of treatment with systemic antipsoriatics:

1. Effectiveness in clinical practice ("real world")
2. Benefits and needs on the patients' side
3. Effectiveness in a long-term course over years
4. Optimal maintenance dosages
5. Safety and side-effects profile under routine conditions
6. Use in case of and effect on co-morbidity
7. Reliable predictors of response
8. Benefit and effectiveness of possible combination therapies or alternating use of biologics and systemic therapies

Methods: The registry evaluates the long-term course of 3,500 patients with Pso and PsA treated with systemic antipsoriatics.The registry started for seven treatment arms: Fumaric acid, methotrexate, ciclosporin A, efalizumab, etanercept, infliximab and adalimumab. While efalizumab was withdrawn from the market, ustekinumab was included after authorization. Patients are included at first initiation of a given treatment and will remain in the registry for 5 years, regardless of subsequent therapy. Nationwide, dermatologic practices and hospital ambulances with expertise in systemic and biologic treatment consecutively enrol patients. Follow-ups will be every 3 to 6 months, comprising patient and treatment characteristics, clinical parameters, patient-defined benefit, quality of life and adverse events. Standardized questionnaires will be addressed to the patient and to the dermatologist 12 times at the dermatologic centres. In interim intervals, patients are directly contacted another 9 times by mail. PsoBest is member of the ENCePP network of psoriasis-registries (www.psonet.eu).

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosis of plaque-type psoriasis or psoriasis arthritis confirmed by a dermatologist
* age ≥ 18 years
* being administered a specific systemic drug for the first time
* informed consent to participate
* sufficient language skills (German)

Exclusion criteria:

* lack of informed consent
* patients being participants of clinical trials at the day of admission to the registry (if a patient is included into a clinical trial during the registry follow-ups, the patient data will be recorded, but analysed separately)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with plaque-type psoriasis or psoriatic-arthritis starting the first systemic treatment with authorized atipsoriatic drugs in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2008-01; Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area Severity Index (PASI) | every 6 month for 10 years
  To evaluate clinical outcome of patients exposed to conventional systemic or biologic therapy for psoriasis/psoriatic-arthritis

SECONDARY OUTCOMES:
Dermatology Life Quality Index (DLQI) | every 3 month for 10 years
  To evaluate disease related quality of life of patients exposed to conventional systemic or biologic therapy for psoriasis/psoriatic-arthritis

OTHER OUTCOMES:
Adverse and serious adverse events | 6 month
  Risk for adverse events and serious adverse events for patients exposed to conventional systemic or biologic therapy for psoriasis/psoriatic-arthritis
Patient Benefit Index (PBI) | every 3 months for 10 years
  To evaluate the patient benefit of conventional systemic or biologic therapy for psoriasis/psoriatic-arthritis
EuroQol Questionnaire (EQ-5D) | every 3 months for 10 years
  To evaluate general state of health of patients exposed to conventional systemic or biologic therapy for psoriasis/psoriatic-arthritis
Questionnaire on Supply Quality in Dermatology (FVQ-d) | every 3 months for 10 years
  To evaluate care characteristics of conventional systemic or biologic therapy for psoriasis/psoriatic-arthritis
Health Assessment Questionnaire (HAQ) | every 6 months for 10 years
  To evaluate arthritis severity of patients exposed to conventional systemic or biologic therapy for psoriasis/psoriatic-arthritis
Patient Global Assessment (Skin: PaGAs, Arthritis: PaGAa) | every 3 months for 10 years
  To evaluate global severity of skin and arthritis in patients exposed to conventional systemic or biologic therapy for psoriasis/psoriatic-arthritis
Physician Global Assessment (Skin: PGAs, Arthritis: PGAa) | every 6 months for 10 years
  To evaluate global severity of skin and arthritis in patients exposed to conventional systemic or biologic therapy for psoriasis/psoriatic-arthritis
Disease Activity Score 28 (DAS 28), American College of Rheumatology Score (ACR20), Psoriatic Arthritic Response Criteria (PsARC) | every 6 months for 10 years
  To evaluate arthritis severity of patients exposed to conventional systemic or biologic therapy for psoriasis/psoriatic-arthritis

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Augustin, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Nationwide group of dermatological centers, hospitals and medical offices, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: PsoBest - the German psoriasis registry — https://www.psobest.de/
- See also: German Center for Health Services Research in Dermatology — https://www.uke.de/kliniken-institute/institute/versorgungsforschung-in-der-dermatologie-und-bei-pflegeberufen/index.html
- See also: PsoNet - the European registry of psoriasis — https://catalogues.ema.europa.eu/network/25161
- See also: Swiss Dermatology Network for Targeted Therapies (SDNTT) — https://www.sdntt.ch/de/